CLINICAL TRIAL: NCT02645266
Title: Mean Visual Acuity Changes Following Five Injections of Aflibercept and the Relationship Between Ocular and Serum Cytokine Levels and Mean Visual Acuity Gains in DME Patients
Brief Title: Mean Visual Acuity Changes Following Five Injections of Aflibercept
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHC-RD-SOP-038
Record Dates: First submitted 2015-12-30; First posted 2016-01-01 (Estimated); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aflibercept Injection [Eylea] group (Experimental): Intervention: Subjects will be receiving a (2mg/ml) dose of VEGF-Trap, injected intravitreally at the start of every month, for the 4 months duration of the trial.
  Interventions: Drug: Aflibercept Injection [Eylea]

INTERVENTIONS:
Drug: Aflibercept Injection [Eylea] — Subjects will be administered 2.0mg Aflibercept intraocular injection each month for 5 consecutive months. After the 5th month, the serum cytokine levels in blood work will be assessed as well as patients's visual acuity, and eye pressures. Upon completion of the trial, patients will resume receiving the usual standard of care.
  Other Names: Eylea treatment

SUMMARY:
Diabetic Macular Edema is a serious ocular consequence of poorly controlled diabetes. Even though significant research has been done to clarify the pathogenesis of DME, a clear causal pathway of the complication is of yet undetermined. However, there is some consensus among researchers that a cascade of inflammatory markers plays an important role in the disease process. The study hopes to better delineate the role these inflammatory markers play by investigating whether basal levels predict response or lack thereof to Aflibercept.

DETAILED DESCRIPTION:
Diabetic macular edema (DME) is a common and serious complication of diabetic retinopathy and is one of the leading causes of vision loss in the developed world. Traditionally, DME was treated with focal grid laser which was not very efficacious. More recently, over the last decade, the development of intravitreal steroids such as Triamcinolone acetonide and anti- vascular endothelial growth factor antibodies such as Bevacizumab (off label usage), Ranibizumab and Aflibercept have proven to be promising. In fact, Aflibercept, being the latest anti-VEGF entering the market, was found superior to traditional treatment in DA VINCI, VIVID DME and VISTA DME studies and there are more trials ongoing. Also, several trials have shown steroids to be superior to laser treatments. The steroids continue to have a role in management of patient refractory to other treatments. This is thought to be due to the inflammatory nature of diabetic macular edema.

Much of the recent success in treatment of DME is owed to the recent developments in our understanding of the inflammatory cascade in a diabetic eye specially the discovery and therapeutic targeting of VEGF. The pathophysiology of DME is thought to be complex and is yet to be fully elucidated; however, a review of literature reveals that there is consensus amongst researchers and clinicians with regards to the importance of disruption of blood retinal barrier involving numerous inflammatory mediators and cytokines in this process. It has been shown that the interruption in BRB is not merely a direct consequence of hyperglycemia but the outcome of inflammatory cascade initiated by chronic hyperglycemia. Chronic hyperglycemia leads to increased production of pro-inflammatory molecules such as advanced glycation end products (AGEs) which are molecules that promote formation of abnormal cross-links in between proteins. These compounds in turn lead to disruptions of the functioning BRB through the up regulation of several inflammatory pathways. Currently the best method to battle AGEs is to prevent their formation through tight glycemic control and the development of therapies has been focused on targeting downstream inflammatory and angiogenic mediators such as VEGFs. It has been shown that VEGFs( VEGF A, B, C, D, E and PLGF) play a major role in neovascularization, formation of new highly friable blood vessels, increased permeability and disruption of BRB with VEGF-A being the most potent promoter of neovascularization. Other factors involved include pigment epithelial derived factor (PEDF), Interleukin-6 and 8( IL-6 and 8), monocyte chemotactic protein-1 (MCP-1), Interferon gamma protein 10(IP-10) etc. It is theorized that some factors play a protective role against the pathogenesis of DME, including PEDF, FLT3L, GM-CSF, IP-10, IFN alpha. It is therefore the lack of balance of these factors that is thought to play a major role in diabetic eye disease.

Since, not all patients respond to anti-VEGF therapies injections; researchers have been pursuing other cytokines and inflammatory mediators as the culprit in the non-responsive group. Up-to-date there have been numerous studies investigating the levels of cytokines in the eyes of diabetic patients and based on our extensive review of the literature this/these mystery molecules can be any of the following cytokines: IL-1, IL-6, IL-7, IL-8, IL-10, IL-12, MCP-1, MCP-3, IP-10,VEGF, PLGF, PEDF, ICAM-1, VCAM-1, GM-CSF, GRO(CXCL-1), TNF-alpha, TGF- beta, Eotaxin, FGF-2, FLT3L,IFN alpha, MDC, MIG(CXCL 9), PKC, and MMP-9. These cytokines may also present a novel path to monitor disease activity.

Until now, there has not been a study attempting to determine whether basal cytokine levels are an indication to response to treatment or lack thereof. It is therefore, in our opinion, essential to carry out such a study as a significant relationship between (an) elevated/ suppressed cytokine and letters gained on best corrected visual acuity or a relationship between an elevated cytokine and not responding to our VEGF treatments could present a path for deciding whether a patient is suited for the anti-VEGF treatment at hand. In addition, it could pave the way for development of a new medication that could act complementary to our current treatments. Above all, we hope to assist eye surgeons and physicians to help their patients with the treatment that fits them the best.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of DME by a retina specialist
2. Age: 18 or older
3. VA between 25 and 75 letters at baseline
4. Treatment naïve

Exclusion Criteria:

1. Unwilling to sign consent form
2. Previous anti-VEGF intravitreal treatment in affected eye
3. Actively taking systemic steroids
4. Ocular inflammatory disease or autoimmune disease
5. Previous laser treatment for DME within last 3 months .
6. Any ocular surgery within the last 3 months.
7. Previous retina surgery( PPV, ERM surgery etc)
8. Medically uncontrolled glaucoma
9. Any other retinal condition( CRAO, CRVO, wAMD, geographic atrophy)
10. Individuals with disabilities that prevent accurate vision testing
11. Proliferative diabetic retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To determine change in BCVA from baseline to month 5 of aflibercept treatment | 5 months
  To determine mean visual acuity letters gain following 4 injections Aflibercept compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada